CLINICAL TRIAL: NCT06189144
Title: Testing the Effectiveness of an Intervention in Irritative Contact Dermatitis:Randomized Controlled Trial
Brief Title: Testing an Intervention in Irritative Contact Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Dario Leskur, assistant professor, University of Split, School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 2181-L98-03-04-23-0030
Record Dates: First submitted 2023-09-13; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Contact Dermatitis; Contact Dermatitis Irritant
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Irritant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): SLS irritation model and Treatment
  Interventions: Other: Emollient cream treatment
- placebo comparator (Placebo Comparator): SLS irritation model and No Treatment
  Interventions: Other: no treatment

INTERVENTIONS:
Other: Emollient cream treatment — Rilastil Difesa Sterile cream
  Arms: experimental arm
Other: no treatment — no treatment
  Arms: placebo comparator

SUMMARY:
An eczematous reaction is an inflammatory intolerance response of the skin. In acute phase the reaction is characterized by erythema and blistering while in the chronic phase it presents as dryness, itchiness and lichenification. Irritative contact dermatitis describes these patterns of reaction in response to toxicity of chemicals on the skin cells, which trigger inflammation by activation of the innate immune system.

DETAILED DESCRIPTION:
An eczematous reaction is an inflammatory intolerance response of the skin. In acute phase the reaction is characterized by erythema and blistering while in the chronic phase it presents as dryness, itchiness and lichenification. Irritative contact dermatitis describes these patterns of reaction in response to toxicity of chemicals on the skin cells, which trigger inflammation by activation of the innate immune system. Therefore, the aim of this study was to see if omega cream, as proposed by its mechanism of action, could improve SLS induced contact dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers who gave written informed consent

Exclusion Criteria:

* · skin cancer

  * skin disease
  * skin damage on measurement sites
  * use of corticosteroids, antihistamines and immunomodulators a month prior the inclusion and during the trial
  * use of drugs that may cause photosensitivity
  * use of emollients three days prior the inclusion in the trial
  * non-adherence to the trial protocol
  * exposure to artificial and excessive natural ultraviolet (UV) radiation
  * pregnancy and lactation
  * history of vitiligo, melasma and other pigmentation and photosensitivity disorders
  * immunosuppression
  * allergic or irritant reactions to the constituents of the cream

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
TEWL measurement with Khazaka probe | through study completion, an average of 1 year
  Transepidermal water loss
hydration measurement with corneometer probe | through study completion, an average of 1 year
  corneometer assessed stratum corneum hydration level
erythema measured with mexameter | through study completion, an average of 1 year
  mexameter assessed redness

SECONDARY OUTCOMES:
clinical score according to dermatologist scale | through study completion, an average of 1 year
  Skin response to irritation and treatment will be assessed using a five-point scale to describe changes in skin erythema, roughness, scaling, oedema, and fissure

CONTACTS AND LOCATIONS:
Overall Officials: josipa bukic, Study Chair — University of Split, School of Medicine
Locations (1):
- School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: ICF, CSR
Time Frame: On request
Access Criteria: On request